CLINICAL TRIAL: NCT03054714
Title: Prospective, Randomized Study of Long-term Hemodialysis Catheter Removal, Versus Guidewire Exchange to Treat Catheter Related Blood Stream Infection
Brief Title: Long-term Hemodialysis Catheter Removal and Delayed Replacement, Versus Exchange Over a Guidewire to Treat Catheter Related Blood Stream Infection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Hossam M. Saleh, Assistant Prof. of vascular surgery, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: tunneled hemodialysis
Record Dates: First submitted 2017-02-10; First posted 2017-02-16 (Actual); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Catheter Related Blood Stream Infection

STUDY DESIGN:
Who Masked: Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group A (Active Comparator): exchange of the infected catheter with a new one over a guidewire
  Interventions: Device: catheter replacement
- group B (Active Comparator): removal of the infected catheter followed by delayed placement of a new catheter 3 to 10 days later
  Interventions: Device: catheter replacement

INTERVENTIONS:
Device: catheter replacement — catheter removal and delayed replacement, versus exchange over a guidewire

SUMMARY:
Prospective, randomized Study of tunneled cuffed hemodialysis catheter removal and delayed replacement, versus exchange over a guidewire to treat catheter related blood stream infection

DETAILED DESCRIPTION:
The aim of this study was to compare the clinical outcomes of catheter-related (CRBSI) managed with two different strategies: Guidewire exchange of the infected catheter with a new one over a guidewire versus catheter removal with delayed replacement.

ELIGIBILITY:
Inclusion Criteria:

* All patients end stage renal disease on hemodialysis from tunneled cuffed dialysis catheters with suspected catheter-related bloodstream infection with no identifiable infection source except the catheter were included.

Exclusion Criteria:

* metastatic infection,

Ages: 14 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 798 (Actual)
Dates: Start 2011-11-01 (Actual); Primary Completion 2016-11-30 (Actual); Study Completion 2016-11-30 (Actual)

PRIMARY OUTCOMES:
infection free survival | 45 days

REFERENCES:
- [Derived] Almeida BM, Moreno DH, Vasconcelos V, Cacione DG. Interventions for treating catheter-related bloodstream infections in people receiving maintenance haemodialysis. Cochrane Database Syst Rev. 2022 Apr 1;4(4):CD013554. doi: 10.1002/14651858.CD013554.pub2. PMID 35363884